CLINICAL TRIAL: NCT06879730
Title: Retrospective Evaluation of Minimally-Invasive Surgical Strategies in Ovarian Neoplasms (REMISSION Study)
Acronym: REMISSION
Status: Recruiting | Type: Observational
Sponsor: Jvan Casarin, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Jvan Casarin, MD PhD, Associate Professor of Obstetrics and Gynecology Director, Research Center for Gynecologic Oncology and Minimally Invasive Surgery, University of Insubria, OB/GYN Consultant, Università degli Studi dell'Insubria
Organization: Università degli Studi dell'Insubria (Other)
Other Study IDs: 55/2024
Record Dates: First submitted 2024-12-01; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-12

CONDITIONS: Early-stage Epithelial Ovarian Cancer
Keywords: early-stage epithelial ovarian cancer; minimally invasive surgery
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients treated with minimally invasive approach
- Patients treated with open surgery

SUMMARY:
This observational study aims to evaluate the outcomes of patients with early-stage epithelial ovarian cancer who are treated with minimally invasive surgery (such as laparoscopic or robotic surgery). Specifically, the study will look at:

1. Post-Surgery Complications

   * What is the rate of complications within 30 days after surgery?
   * How often do patients require readmission to the hospital, re-operation, or conversion to open surgery?
2. Cancer Outcomes

   * What is the rate of cancer upstaging (when the cancer spreads to a more advanced stage during surgery for example because of an intra-operative ovarian cyst rupture)?
   * What are the overall survival and disease-free survival rates for patients treated with minimally invasive surgery?

Researchers will compare two groups of patients:

Group 1: Patients with early-stage ovarian cancer treated with minimally invasive surgery.

Group 2: Patients with early-stage ovarian cancer treated with open surgery. The goal is to see if there are any differences in post-surgery complications, recovery, and cancer outcomes between the two groups.

Fertility-Sparing Treatment:

The study will also compare patients who are undergoing fertility-sparing treatments for early-stage ovarian cancer. Two subgroups will be looked at:

* Patients receiving fertility-sparing surgery through a minimally invasive procedure.
* Patients receiving fertility-sparing surgery through an open surgery. The same outcomes (complications, survival, etc.) will be assessed and compared between these two groups as well.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with apparent early-stage epithelial ovarian cancer at preoperative evaluation
2. Patients who underwent surgery between January 2014 and December 2023
3. Patients who underwent open or minimally invasive surgical staging (Laparoscopic or Robotic-assisted approach) or restaging procedure
4. Patients with final pathology report of Epithelial Ovarian Cancer

Exclusion Criteria:

1. Patients who have not performed a complete surgical staging
2. Patients who underwent neoadjuvant chemotherapy
3. Patients with invasive synchronous tumor
4. Patients with no informed consent
5. Patients with ASA class score of 4 or 5

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — patients eligible need to have apparent early stage epithelial ovarian cancer, therefore they need to have a female reproductive system
Study Population: The current study is a retrospective multicentric international observational study of data from patients with apparent early-stage epithelial ovarian cancer who underwent minimally-invasive or open surgery between January 2014 and December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To assess the number of patients with 30-day post-operative complication in the two groups (minimally invasive surgery and open surgery) | From surgery to post-operative day 30
To assess the number of patients with 30-day post-operative hospital readmission in the two groups (minimally invasive surgery and open surgery) | From surgery to post-operative day 30
To assess the number of patients with 30-day post-operative reoperation in the two groups (minimally invasive surgery and open surgery) | From surgery to post-operative day 30
To assess the rate of upstaging in the two groups (minimally invasive surgery and open surgery) | At the time of surgery
To assess the rate of conversion in the minimally invasive surgery group | At the time of surgery

SECONDARY OUTCOMES:
To analyze predictor of recurrence and oncological outcomes in terms of disease-free survival (DFS) and overall survival (OS) in the minimally invasive surgery and in the open surgery groups | From the date of surgery to the date of the last follow-up or the date of recurrence/death, whichever occurs first, assessed up to 300 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Filippo del Ponte, Varese, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided